CLINICAL TRIAL: NCT02297789
Title: Evaluation of a Full Face Mask and Headgear for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIA-152
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Headgear 1 (Experimental): Full Face Mask with Headgear 1
  Interventions: Device: Investigative Full Face Mask with Headgear
- Headgear 2 (Experimental): Full Face Mask with Headgear 2
  Interventions: Device: Investigative Full Face Mask with Headgear

INTERVENTIONS:
Device: Investigative Full Face Mask with Headgear

SUMMARY:
Currently Fisher & Paykel Healthcare (FPH) is developing a new full face mask. The objective of this clinical investigation is to evaluate the usability and acceptance of the investigative mask, the effectiveness of the seal and headgear.

The participant will be randomised to use either full face mask prototype 1 or 2 as according to the randomization log for 7 ± 3 days in home. The participant will then crossover to the other full face mask prototype to use in home for 7 ± 3 days. Neither the investigators or the participants will be blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* AHI ≥ 5 from the diagnostic night
* ≥ 18 years of age
* Either prescribed APAP or CPAP or Bi level for OSA
* Existing full face users

Exclusion Criteria:

* Inability to give informed consent
* Participant intolerance to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or CO2 retention
* Pregnant or think they may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The mask is comfortable and is effective for the participant during in-home use | 1 week for each mask prototype in-home
  Performance in relations to leak and comfort of each prototype and how it compares to their usual mask, as measured by a custom questionnaire, daily participant feedback log and PAP device data.

SECONDARY OUTCOMES:
Acceptability of the Full Face mask prototypes | 1 week for each mask prototype in-home
  Preference for one of the Full Face Mask prototypes design through a custom questionnaire and a daily participant feedback log

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, BSc, Principal Investigator — Fisher & Paykel Healthcare
Locations (1):
- Fisher & Paykel Healthcare Ltd., Auckland, East Tamaki, New Zealand